CLINICAL TRIAL: NCT02264379
Title: Effectiveness and Toxicity of a Percutaneous High-dose Radiotherapy in Patients With Oligometastases of Prostate Carcinoma
Brief Title: Percutaneous High-dose Radiotherapy in Patients With Oligometastases of Prostate Carcinoma
Acronym: Oli-P
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Tobias Hölscher, Dr., Technische Universität Dresden
Other Study IDs: STR - Oli-P - 2014
Record Dates: First submitted 2014-05-22; First posted 2014-10-15 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Oligometastatic Disease; Prostate Cancer
Keywords: Oligometastatic Disease; Prostate Cancer; Stereotactic Radiotherapy; androgensensitive
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood before therapy, at the end of radiotherapy, three months after the end of radiotherapy and at progress before starting further treatment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal fractionated irradiation
  Interventions: Radiation: normal fractionated irradiation
- hypo fractionated irradiation
  Interventions: Radiation: hypo fractionated irradiation

INTERVENTIONS:
Radiation: normal fractionated irradiation — 25*2 Gy (once a day, 5 days a week)
  Groups: normal fractionated irradiation
Radiation: hypo fractionated irradiation — 3*10 Gy (once a day, 2-3 days a week)
  Groups: hypo fractionated irradiation

SUMMARY:
The purpose of this study is to evaluate the outcomes of patients treated with an high dose radiation regimen using either stereotactic hypofractionated or normofractionated radiotherapy for oligometastatic prostate cancer and to establish efficacy (producing a desired result or effect) and safety in this setting.

DETAILED DESCRIPTION:
Study Groups:

If the patient found to be eligible to take part in this study, the patient will be assigned to a study group based on the size of the lesion(s) and the discretion of the responsible physician. Up to 71 patients will be enrolled in the study.

If the patient is treated with standard radiotherapy, the patient will receive 25 fractions of 2 Gy to the metastases, the treatment duration will be 5 weeks.

If the patient is treated with image-guided hypofractionated radiotherapy, the patient will receive 3 fractions of 10 Gy to the metastases, the treatment duration will be 1 week.

Radiation Planning and Treatment:

During all radiation treatments, the images that are taken during the treatment will be closely analyzed after treatment is over. The patient will have 3 to 25 radiation treatments per metastasis depending on the discretion of the responsible physician.

The rest of the radiation treatment planning and treatment delivery appointments will be unchanged. The dose given to the tumor and number of treatments the patient will receive, will be determined by the discretion of the responsible physician, and is not affected by taking part in this study.

Follow-Up Visits:

After the radiation treatment schedule ends, the patient will return for follow-up visits at the following time points:

* At 3 months
* Then, every 3 months for 1 year, and then
* 1 time a year after that, for as long as possible Additional follow up visits may be scheduled, if the responsible physician thinks they are needed.

At these visits, the following tests and procedures will be performed:

* Any updates to the medical history of the patient will be recorded and the patient will be asked about any side effects the patient may be having.
* The patient's performance status will be recorded.
* The patient's complete symptom questionnaires will be reviewed.
* The patient will have a clinical examination
* The patient will have follow-up imaging (such as an MRI) to check the status of the disease.

This is an observational study. Radiation therapy is delivered using CE-certified and commercially available methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient with good general condition (WHO 0-1)
* No comorbidities which limit the further life expectancy of the patient to <5 years (opinion of the physician)
* Histologically confirmed prostate cancer
* State after definitive local therapy, such as radical prostatectomy or definitive radiotherapy (even after neo-/-adjuvant hormone therapy, after postoperative radiotherapy)
* PSA relapse after primary therapy or radiological unique metastasis, present complete staging (up to 8 weeks old) by CT thorax/ abdomen/ pelvis and bone scan alternatively a hybrid imaging PET (positron emission tomography) (acetate PET, PET-PSMA, NAFL-PET) and CT / MRI is sufficient
* Imaging detection of individual metastases (up to 5, depending on the situation) that a Radiation therapy are available (histological confirmation of the MET is not required)
* No parallel participation to further clinical therapeutic trials to 4 weeks and after radiation
* Consent of the patient and written informed consent

Exclusion Criteria:

* severe comorbidity which limit the further life expectancy of the patient to <5 years (opinion of the physician)
* PSA in PSA relapse> 10ng/ml
* Ongoing androgen deprivation at the time of study inclusion
* not been carried out local therapy
* no histological confirmation of prostate cancer
* lack of compliance
* absence of consent of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oligometastases (1-5) and state after local therapy of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Late Toxicity at year 2 after ablatvie radiotherapy | 24 months after therapy
  The toxicity will be scored (CTCAE 4.03) at each follow up visit, the status will be recorded by clinical examination and radiological imaging.

SECONDARY OUTCOMES:
Early toxicity | until day 90 after start radiotherapy
  The toxicity will be scored (CTCAE 4.03) at 3 months follow up visit, the status will be recorded by clinical examination and radiological imaging.
Quality of life (QLQ-C30 and QLQ-PR25) during Follow-up | 24 months after end of therapy
  QoL will be assessed with the QoL-Questionaires QLQ-C30 and QLQ-PR25 at baseline, 3, 12 and 24 months after treatment.
Local control of irradiated tumor manifestations | 24 months after end of therapy
  The tumor response will be evaluated (RECIST) at follow up visit 3,12 and 24 months after end of treatment, the status will be recorded by clinical examination and radiological imaging.
Therapy-free survival | 24 months after end of therapy
  Therapy-free survival will be assessed as time from start of radiation to start of systemic treatment or androgen deprivation. The status will be assessed at each follow-up visit.
PSA relapse-free survival | 24 months after end of therapy
  PSA relapse-free survival will be assessed as time from start of radiation to PSA-rise more than 20% above baseline. PSA - value will be assessed by blood testing.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hölscher, Dr., Principal Investigator — Technische Universität Dresden, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology
Locations (2):
- Germany (2):
  - Technische Universität Dresden, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, Dresden, Saxony
  - Universitätsklinikum Tübingen, Department of Radiation Therapy and Radiation Oncology, Tübingen

IPD SHARING:
Plan to Share IPD: No